CLINICAL TRIAL: NCT06990893
Title: Comparison of the Analgesic Effect of Oliceridine Versus Morphine or Sufentanil for Postoperative Analgesia in Lumbar Surgeries: a Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sun Ling
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-10

CONDITIONS: Sufentanil; Morphine; Validity; Safety; Oliceridine
Keywords: Sufentanil; Safety; Morphine; oliceridine
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Morphine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The oliceridine group(A) (Experimental): A loading dose of 1.5mg of oliceridine was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.01 mg.kg-1.h-1 orselidine was connected and diluted with normal saline to 100ml at a rate of 2ml per hour
  Interventions: Drug: Oliceridine
- The morphine group(M) (Experimental): A loading dose of 4mg of morphine was intravenously injected. Ten minutes later, an intravenous analgesic pump was connected to 0.03mg.kg-1.h-1 morphine mixed with normal saline to 100ml at a rate of 2ml per hour
  Interventions: Drug: Morphine
- The sufentanil group(S) (Experimental): A loading dose of 4ug of sufentanil was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.03ug.kg-1.h-1 was connected. Sufentanil was mixed with normal saline to 100ml at a rate of 2ml per hour
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Oliceridine — a loading dose of 1.5 mg of oliceridine was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.01 mg.kg-1.h-1 oliceridine was connected with normal saline to 100 ml at a rate of 2 ml per hour
  Arms: The oliceridine group(A)
Drug: Morphine — a loading dose of 4 mg of morphine was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.03 mg.kg-1.h-1 morphine was connected with normal saline to 100 ml at a rate of 2 ml per hour
  Arms: The morphine group(M)
Drug: Sufentanil — A 4 ug loading dose of sufentanil was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.03 ug.kg-1 h-1 was connected. sufentanil was mixed with normal saline to 100 ml at a rate of 2 ml per hour
  Arms: The sufentanil group(S)

SUMMARY:
Objective: To compare the application of oxelidine in postoperative analgesia after orthopedic lumbar spine surgery with morphine or sufentanil, and to explore the efficacy and safety of postoperative analgesia.

Method: Researchers included 90 patients with American Society of Anesthesiologists (ASA) physical conditions I and III, aged 18 to 65 years, who were scheduled to undergo orthopedic lumbar general anesthesia surgery at an appropriate time. The patients were randomly divided into 3 groups, with 30 cases in each group: The oxeridine group (Group A), where a loading dose of 1.5mg of oxeridine was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.01mg/kg-1.h-1 was connected. Oxeridine was mixed with normal saline to 100ml at a rate of 2ml/h. Morphine group (Group M), a loading dose of 4mg of morphine was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.03mg.kg-1.h-1 morphine was connected with normal saline to 100ml at a rate of 2ml/h. Sufentanil group (Group S), a 4u loading dose of sufentanil was intravenously injected. Ten minutes later, an intravenous analgesic pump of 0.03ug.kg-1.h-1 was connected. Sufentanil was combined with normal saline to 100ml at a rate of 2ml/h.The resting and exercise VAS pain scores of the three groups of patients at 30 minutes, 2 hours, 6 hours, 12 hours, 24 hours and 48 hours after the operation and adverse reactions within 48 hours were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spine surgery with ASA grades I-III
* Aged 18-65 years
* Ethically, the patient voluntarily accepted this trial and signed the informed consent form

Exclusion Criteria:

* Severe respiratory and circulatory system diseases
* Nervous system disease
* Mental and psychological disorders
* Abnormal liver and kidney functions
* Participated in another drug clinical research within the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The VAS pain scores at rest and during exercise of the three groups of patients after the operation | at 30 minutes, 2 hours, 6 hours, 12 hours, 24 hours and 48 hours after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China

IPD SHARING:
Plan to Share IPD: No